CLINICAL TRIAL: NCT06691854
Title: The Effect of the Intrapartum Care Model Given in Line With the World Health Organization (WHO) Recommendations on Women's Perception of Respectful Maternity Care, Birth Experiences and Perception of Traumatic Birth.
Brief Title: Women's Perception of Respectful Maternity Care, Birth Experiences and Perception of Traumatic Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Assoc. Prof. Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/982
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Maternity; Birth, First; Traumatic Birth; Intrapartum Fetal Distress
Keywords: Respectful maternity care scale; Birth experience scale; Traumatic birth perception scale; WHO Intrapartum Care Recommendations
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (No Intervention): Pregnant women who apply to the hospital for delivery, have a cervical dilatation of 5 cm or more, agree to participate in the study and are assigned to the control group;
  * A personal information form will be applied at the first clinic admission.
  * Pregnant women assigned to the control group will receive routine intrapartum care provided at the hospital.
  * The labor process of the pregnant woman will be recorded on the birth experience monitoring form.
  * The mother and baby will receive routine postpartum care provided at the hospital.
  * After delivery, the Respectful maternity care scale, Birth experience scale, Traumatic birth perception scale will be applied.
- The group that applied the Intrapartum Care Model (Experimental): Pregnant women who apply to the hospital for delivery, have cervical dilatation of 5 cm and above, agree to participate in the study and are assigned to the intervention group;
  * A Personal Information form will be applied at the first clinic admission.
  * All primiparous pregnant women assigned to the intervention group will be applied the intrapartum care model by the research midwife during the labor process and after birth in line with the WHO positive birth recommendations (Table 1).
  * The labor process of the pregnant woman will be recorded on the birth experience follow-up form.
  * After birth, the Respectful maternity care scale, Birth experience scale, Traumatic birth perception scale will be applied.
  Interventions: Other: The group that applied the Intrapartum Care Model

INTERVENTIONS:
Other: The group that applied the Intrapartum Care Model — Pregnant women who apply to the hospital for delivery, have cervical dilatation of 5 cm and above, agree to participate in the study and are assigned to the intervention group;
  A Personal Information form will be applied at the first clinic admission. All primiparous pregnant women assigned to the intervention group will be applied the intrapartum care model by the research midwife during the labor process and after birth in line with the WHO positive birth recommendations.
  The labor process of the pregnant woman will be recorded on the birth experience follow-up form.
  After birth, the Respectful maternity care scale, Birth experience scale, Traumatic birth perception scale will be applied.
  Arms: The group that applied the Intrapartum Care Model

SUMMARY:
The effect of the ıntrapartum care model given in line with the world health organization (WHO) recommendations on women's perception of respectful maternity care, birth experiences and perception of traumatic birth

DETAILED DESCRIPTION:
The research is a randomized controlled trial. The research will conducted with 124 primiparous pregnant women (intervention group n=62, control group n=62) who were hospitalized in the delivery unit of Aksaray Training and Research Hospital between September 2023 and January 2024. The pregnant women in the intervention group will given the intrapartum care model in line with WHO recommendations after cervical dilation reached 5 cm. The control group will received only the standard intrapartum care in the hospital. Data will be collected using the personal information form, birth follow-up form, respectful maternal care scale, birth experience scale, and traumatic birth perception scale.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years of age or older,
* Those who are in term pregnancy (38-41 weeks),
* Those who are primiparous,
* Those who have a single, healthy, vertex positioned fetus,
* Those who have cervical dilatation of 5 cm or more,
* Those who can speak and understand Turkish,
* Those who voluntarily agree to participate in the research.

Exclusion Criteria:

* Those with chronic diseases (hypertension, diabetes, etc.),
* Those with a diagnosed mental illness (depression, anxiety or other psychotic disorder, etc.),
* Those with maternal and fetal complications (oligohydramnios and polyhydramnios, placenta previa, preeclampsia, premature membrane rupture, presentation anomalies, intrauterine growth retardation, fetal anomalies, intrauterine death, macrosomic baby, cord prolapse, etc.),
* Those with any complications that prevent vaginal birth (cephalopelvic disproportion, etc.),
* Elective cesarean section,
* Those who became pregnant with assisted reproductive techniques,
* Those who received childbirth preparation training.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of sociodemographic characteristics of pregnant women before the intervention with the questionnaire | 6 months
  Sociodemographic of pregnant women will be collected through surveys and compared and reported
Comparison of pre-intervention obstetric characteristics of pregnant women with a questionnaire | 6 months
  Obstetric of pregnant women will be collected through surveys and compared and reported
Comparison of the delivery times of pregnant women through a survey | 6 months
  The duration of labor of the groups will be collected through surveys and compared and reported
Comparison of the means of the respectful birth care scale among pregnant women by group | 6 months
  The respectful maternity care scale will be applied to pregnant women. The respectful maternity care scale is 19-95 points (min-max), and as the score increases, women's respectful maternity care increases.
Comparison of the means of the birth experience scale among pregnant women by group | 6 months
  The birth experience scale will be applied to pregnant women. The birth experience scale is 22-88 points (min-max), and as the score increases, it indicates that the expectant mother has a good birth experience.
Comparison of the means of the traumatic birth perception scale among pregnant women by group | 6 months
  The traumatic birth perception scale will be applied to pregnant women. The traumatic birth perception scale is 0-130 points (min-max). The scale shows that the 0-26 point range is "very low", the 27-52 point range is "low", the 53-78 point range is "medium", the 79-104 point range is "high", and the 105-130 point range is "very high" traumatic birth perception level.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çankaya, PhD, Principal Investigator — Selcuk University
Locations (1):
- Seyhan Çankaya, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No